CLINICAL TRIAL: NCT04652492
Title: A Multicentric, Open-Label Study to Evaluate Tislelizumab in Combination With Transarterial Chemoembolization as First-Line Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Tislelizumab in Combination With TACE in Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dr., Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-2004-IIT
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: TACE; tislelizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab in combination with cTACE (Experimental): Tislelizumab in combination with on-demanded cTACE
  Interventions: Drug: Tislelizumab in combination with cTACE

INTERVENTIONS:
Drug: Tislelizumab in combination with cTACE — On-demanded cTACE in combined with tislelizumab (200mg q3w ivgtt on day 4 of each 21-day cycle)
  Other Names: BGB-A317

SUMMARY:
A multicentric, open-label, single-arm prospective study to assess the efficacy and safety of tislelizumab combined with TACE as first-line treatment in patients with unresectable BCLC stage C HCC.

DETAILED DESCRIPTION:
This is a multicentric, open-label, single-arm prospective study to assess the efficacy and safety of tislelizumab combined with conventional transarterial chemoembolization(cTACE) as first-line treatment in BCLC stage C HCC patients without extrahepatic spread. The primary endpoint is time to progression (TTP).

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old on the day the patients voluntary to participate in the study and signing in ICF.
2. Histological or clinical diagnosis of HCC.
3. BCLC stage C patients ineligible for surgical resection or liver transplantation.
4. No prior systemic therapy for HCC (including immunotherapy).
5. Have at least one uni-dimensional lesion measurable by CT scan or magnetic resonance imaging per mRECIST.
6. Child-Pugh A-B7.
7. ECOG PS 0-1.
8. Adequate hematological function (absolute neutrophil count ≥ 1.5 X 109/L, platelets count≥50 X109/L, and hemoglobin ≥85 g/L); Adequate hepatic function (both AST and ALT ≤ 3 ULN, serum total bilirubin ≤ 34.2 umol/L or 2mg/dl, serum albumin ≥ 29g/L); Adequate renal function (eGFR > 30 ml/min/1.73 m2)
9. For patients with HBV or HCV infection, HBV DNA less than 500 IU/ml (2500 copies/ml) or HCV RNA detectable.
10. life expectancy of more than 3 months.
11. Patients must be able to understand and willing to sign a written informed consent document.
12. Patients suitable for TACE therapy assessed by investigators.

Exclusion Criteria:

1. Tumor thrombus involving main trunk of portal vein or inferior vena cava.
2. Prior local-regional therapy before beginning of study treatment (surgery or ablation allowed at BCLC stage 0-B) or radiotherapy on liver cancer.
3. Disease history of grade 2 or more hepatic encephalopathy.
4. Extrahepatic metastasis on baseline imaging.
5. HIV infection or syphilis.
6. Prior therapies with any anti-PD-1, anti-PD-L1, anti-PD-L2 or anti-CTLA-4 agents.
7. Tumor diffuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
TTP assessed by independent review committee(IRC) | up to 24 months after enrollment or study close
  Defined as the time from the date of first cTACE to the date of first documentation of disease progression per mRECIST. When pseudoprogression is suspected by investigator, tumor response will be re-assessed per iRECIST to confirm (also applicable for secondary endpoint of efficacy).

SECONDARY OUTCOMES:
TTP assessed by investigators | An expected average of 8 months
  Defined as the time from the treatment initiation to the date of the first objectively documented tumor progression, assessed by investigators per mRECIST.
PFS | An expected average of 8 months
  Defined as the time from the treatment initiation to the date of the first objectively documented tumor progression or death, whichever occurs first, assessed by IRC and investigators, respectively, per mRECIST.
ORR | An expected average of 8 months
  Defined as the proportion of patients with a documented CR or PR, assessed by IRC and investigators, respectively, per mRECIST.
DCR | An expected average of 8 months
  Defined as the proportion of patients whose best overall response (BOR) is CR, PR, or SD, assessed by IRC and investigators, respectively, per mRECIST.
DOR | An expected average of 8 months
  Defined as the time from the first confirmation of objective remission (CR or PR) to the first recording of disease progression or death, whichever occurs first, assessed by IRC and investigators, respectively, per mRECIST.
OS | An expected average of 24 months
  Defined as the time from the treatment initiation to the date of death due to any cause.
Safety | up to 24 months after enrollment or study close
  NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Centre of Interventional Radiology and Vascular Surgery, Department of Radiology, Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No